CLINICAL TRIAL: NCT02396602
Title: miPlan: A Randomized Controlled Trial of miPlan Intervention vs. Standard of Care
Brief Title: miPlan: A Trial of miPlan Intervention vs. Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-0599
Record Dates: First submitted 2015-02-16; First posted 2015-03-24 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Unintended Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): After completing baseline the baseline questionnaire, women randomized to the intervention group will receive an iPad, along with a brief tutorial on iPad navigation, and use the miPlan app for up to 15 minutes. They will complete a post-intervention survey before proceeding to standard of care contraceptive counseling.
  Interventions: Behavioral: miPlan intervention
- Control (No Intervention): After completing baseline the baseline questionnaire, women randomized to the control arm will proceed to standard of care contraceptive counseling.

INTERVENTIONS:
Behavioral: miPlan intervention — miPlan mobile contraceptive counseling waiting room app intervention
  Arms: Intervention

SUMMARY:
Using our experience in digital media, behavior theory, client-centered interventions, and family planning, we have prototyped a digital application ("app")-miPlan-to be used in the clinic waiting room prior to a contraceptive visit. The goal of this research is to refine the app and conduct a randomized controlled trial of the miPlan intervention vs. standard care. The aim of this study is to understand miPlan's impact. The primary outcome is LARC uptake at clinic discharge. The secondary outcomes are contraceptive use at discharge, self-efficacy and decisional balance for highly effective contraception post-app use, contraceptive satisfaction, and intention to continue method use. The research will consist of baseline activities as well as a three-month follow-up call.

DETAILED DESCRIPTION:
Using our experience in digital media, behavior theory, client-centered interventions, and family planning, we have prototyped a digital application ("app")-miPlan-to be used in the clinic waiting room prior to a contraceptive visit. The goal of this research is to refine the app and conduct a randomized controlled trial of the miPlan intervention vs. standard care contraceptive counseling. The aim of this study is to understand miPlan's impact in terms of contraceptive knowledge, intentions and behaviors. The primary outcome is LARC uptake, which will be measured via chart review at clinic discharge, i.e. immediately following a patient's family planning visit. The secondary outcomes are contraceptive use at discharge (measured via chart review immediately following patient's family planning visit), self-efficacy and decisional balance (both measured via adapted validated scales for each) for highly effective contraception post-app use (measured immediately following intervention and prior to contraceptive counseling session), contraceptive satisfaction (measured at 3 months post baseline), and intention to continue method use (measured at 3 months post baseline). The research will consist of baseline activities as well as a three-month follow-up call.

ELIGIBILITY:
Inclusion Criteria:

* African American or Latina female and sexually active with a male partner(s) within the past 6 months,
* age 15 to 29 years
* present for contraception initiation
* English speaking

Exclusion Criteria:

* not currently pregnant or intending pregnancy within the next 6 months
* and not currently using LARC
* not highly intending LARC at enrollment

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
LARC uptake | at time of intervention (baseline (0 weeks)
  uptake of the implant or IUD at time of intervention (measured via contraceptive method choice and delivery by checkbox)

SECONDARY OUTCOMES:
contraceptive use | at time of intervention (baseline (0 weeks))
  use of contraceptive methods at time of intervention (measured via contraceptive method choice and delivery by checkbox)
change in self-efficacy for contraception at 12 weeks | baseline (0 weeks) and 12 weeks
  change in self efficacy for contraceptive method use (measured via validated 5-item attitudinal scale by Galavotti et al 1995) from baseline to 12 weeks
change in decisional balance for highly effective methods at 12 weeks | baseline (0 weeks) and 12 weeks
  change in decisional balance for highly effective methods (measured via validated 10-item attitudinal scale by Galavotti et al 1995) from baseline to 12 weeks
contraceptive satisfaction | 12 weeks post-enrollment
  satisfaction with contraceptive method choice (measured by 4-point Likert scale)
intention to continue method use | 12 weeks post enrollment
  intention to continue contraceptive method use (measured dichotomously)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago, Dept. of OBGYN
Locations (1):
- Planned Parenthood Illinois, Englewood Health Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hebert LE, Hill BJ, Quinn M, Holl JL, Whitaker AK, Gilliam ML. Mobile contraceptive application use in a clinical setting in addition to standard contraceptive counseling: A randomized controlled trial. Contraception. 2018 Oct;98(4):281-287. doi: 10.1016/j.contraception.2018.07.001. Epub 2018 Jul 10. PMID 30006030